CLINICAL TRIAL: NCT01954251
Title: Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A When Co-administered With GSK Biologicals' Seasonal Influenza Vaccine GSK2321138A in Adults Aged 50 Years and Older
Brief Title: Study to Evaluate the Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster Vaccine GSK1437173A When Co-administered With GSK Biologicals' Seasonal Influenza Vaccine GSK2321138A in Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 117036; 2013-000372-15 (EudraCT Number)
Record Dates: First submitted 2013-09-19; First posted 2013-10-01 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-03

CONDITIONS: Herpes Zoster
Keywords: FLU-D-QIV; Adults; Safety; Immunogenicity; co-administration; Herpes zoster
MeSH Terms: conditions — Herpes Zoster

ARMS (2):
- Co-Ad Group (Experimental): The subjects assigned to the Co-Ad group will receive one injection of the FLU-D-QIV vaccine and one injection of the HZ/su study vaccine during the first visit and a second injection of the HZ/su study vaccine during the third visit, two months later.
  Interventions: Biological: Herpes Zoster vaccine GSK 1437173A; Biological: GSK Biologicals' quadrivalent seasonal influenza vaccine FLU-D-QIV GSK2321138A
- Control Group (Active Comparator): The subjects assigned to the Control group will receive all vaccines separately: one injection of the FLU-D-QIV vaccine at the first visit, one injection of the HZ/su study vaccine at the third visit and a second injection of the HZ/su study vaccine at the fourth visit, all two months apart.
  Interventions: Biological: Herpes Zoster vaccine GSK 1437173A; Biological: GSK Biologicals' quadrivalent seasonal influenza vaccine FLU-D-QIV GSK2321138A

INTERVENTIONS:
Biological: Herpes Zoster vaccine GSK 1437173A — 2 doses administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
Biological: GSK Biologicals' quadrivalent seasonal influenza vaccine FLU-D-QIV GSK2321138A — 2 doses administered intramuscularly (IM) in the deltoid region of the dominant arm.
  Other Names: Influsplit™ Tetra (Germany); Fluarix™ Quadrivalent (United States)

SUMMARY:
The purpose of this study is to assess immunogenicity, reactogenicity and safety of GSK Biologicals' HZ/su vaccine when its first dose is co-administered with the FLU-D-QIV vaccine in adults aged 50 years or older compared to administration of vaccines separately.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* A male or female aged 50 years or older, at the time of the first vaccination with the study vaccine(s).
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose (for corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent). A prednisone dose of < 20 mg/day is allowed. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration or planned administration of a vaccine not foreseen by the study protocol within the period starting 30 days before the first dose of study vaccine(s) (HZ/su and/or FLU-D-QIV vaccines) and ending 30 days after the last dose of HZ/su vaccine.
* Administration of an influenza vaccine during the six months preceding entry into the study or planned administration up to the last blood sampling with the exception of the FLU-D-QIV vaccine given during this study.
* Administration of long-acting immune-modifying drugs (e.g. infliximab) within six months prior to the first vaccine dose or expected administration at any time during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination against VZV or HZ and/or planned administration during the study of a VZV or HZ vaccine (including an investigational or non-registered vaccine) other than the study vaccine.
* History of HZ.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, HIV infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of Guillain Barré syndrome.
* Hypersensitivity to latex.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C /100.4°F on rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions before 2 months after the last dose of study vaccine.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Any condition which, in the judgment of the investigator would make intramuscular injection unsafe.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2013-10-03; Primary Completion 2014-06-02 (Actual); Study Completion 2015-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (3):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
- Canada (2):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Toronto, Ontario
- Germany (10):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Dippoldiswalde, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Schwarz TF, Aggarwal N, Moeckesch B, Schenkenberger I, Claeys C, Douha M, Godeaux O, Grupping K, Heineman TC, Fauqued ML, Oostvogels L, Van den Steen P, Lal H. Immunogenicity and Safety of an Adjuvanted Herpes Zoster Subunit Vaccine Coadministered With Seasonal Influenza Vaccine in Adults Aged 50 Years or Older. J Infect Dis. 2017 Dec 12;216(11):1352-1361. doi: 10.1093/infdis/jix481. PMID 29029224
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 117036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 829 subjects enrolled in this trial, 1 subject did not receive vaccination even though subject number had been allocated, hence he/she was excluded from study start.
Groups:
- GSK1437173A + GSK2321138A Group: The subjects assigned to the Co-Ad group received one injection of the FLU-D-QIV vaccine and one injection of the HZ/su study vaccine during the first visit and a second injection of the HZ/su study vaccine during the third visit, two months later.
- Control Group: The subjects assigned to the Control group received all vaccines separately: one injection of the FLU-D-QIV vaccine at the first visit, one injection of the HZ/su study vaccine at the third visit and a second injection of the HZ/su study vaccine at the fourth visit, all two months apart.
Period: Overall Study
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Started | 413 | 415
Completed | 400 | 396
Not Completed | 13 | 19
Not completed — Adverse Event | 5 | 7
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group | Total
Number analyzed (Participants) | 413 | 415 | 828
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (8.3) | 63.4 (8.8) | 63.4 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 218 | 429
  Male | 202 | 197 | 399

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Vaccine Response to Anti-gE Antibodies
Description: The vaccine response(VRR) for anti-gE humoral immunogenicity, as determined by enzyme-linked immunosorbent assay (ELISA),was assessed only in subjects from the GSK1437173A + GSK2321138A Group. The VRR for anti-gE was defined as the percentage of subjects who had at least: a 4-fold increase in the post-dose 2 anti-gE antibody concentration as compared to the pre-vaccination anti-gE antibody concentration, for subjects who were seropositive at baseline (cut-off ≥ 97 mIU/ml), or, a 4-fold increase in the post dose 2 anti-gE antibody concentrations as compared to the anti-gE antibodies cut-off value for seropositivity, for subjects who were seronegative at baseline (cut-off < 97 mIU/ml).
Time Frame: At one month post-dose 2 (Month 3)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity outcome measures were available.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group
Number analyzed (Participants) | 382
Subjects | 366

2. Primary Outcome: Vaccine Response for Anti-gE Humoral Immunogenicity
Description: The vaccine response(VRR) for anti-gE humoral immunogenicity, as determined by enzyme-linked immunosorbent assay (ELISA),was assessed only in subjects from the GSK1437173A + GSK2321138A Group. The VRR for anti-gE was defined as the percentage of subjects who had at least:
  a 4-fold increase in the post-dose 2 anti-gE antibody concentration as compared to the pre-vaccination anti-gE antibody concentration, for subjects who were seropositive at baseline (cut-off ≥ 97 mIU/ml), or, a 4-fold increase in the post dose 2 anti-gE antibody concentrations as compared to the anti-gE antibodies cut-off value for seropositivity, for subjects who were seronegative at baseline (cut-off < 97 mIU/ml).Criterion used: the objective was met if the Lower Limit (LL) of the 95% confidence interval (CI) of the VRR for anti-gE antibody concentrations was at least 60%.
Time Frame: At one month post-dose 2 (Month 3)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GSK1437173A + GSK2321138A Group
Number analyzed (Participants) | 382
Percentage | 95.8 [93.3 to 97.6]

3. Primary Outcome: Adjusted Geometric Mean ELISA Concentrations of Anti-gE Antibodies
Description: Geometric means (GMs) of post-vaccination concentrations (Month 3 for GSK1437173A + GSK2321138A group and Month 5 for Control group) was calculated conditionally to the means of the pre-vaccination log-transformed concentrations for anti-gE (Month 0 for GSK1437173A + GSK2321138A group and Month 2 for Control group). Adjusted Least Squares (LS) means and difference of LS means between the groups were calculated together with 2-sided 95% CIs and back-transformed to the original units to provide GMCs.
Time Frame: At one month post-dose 2 (Month 3 for GSK1437173A + GSK2321138A group and Month 5 for Control group)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 382 | 388
mIU/mL | 52151.6 [48356.0 to 56245.2] | 56247.4 [52177.3 to 60634.9]
Statistical Analysis 1: Comparison: GSK1437173A + GSK2321138A Group vs Control Group; Adjusted ratios of Control group over GSK1437173A + GSK2321138A group in anti-gE antibody ELISA concentrations GMCs at one month after last vaccine dose. An Analysis of Covariance (ANCOVA) model was used to analyse post-vaccination log-transformed concentrations of anti-gE. The fixed-effect model included the minimisation variable (age cohorts) and the treatment as fixed effect. The pre-vaccination log-transformed concentrations were included as continuous covariate; Test type: Non-Inferiority or Equivalence — Comparison at one month after the last dose of HZ/su was performed between the Control group and GSK1437173A + GSK2321138A group. The GSK1437173A + GSK2321138A group was considered as statistically significant non-inferior compared to the Control group in terms of immunogenicity if the UL of the 2-sided 95% CI of the ratio of GMs between the Control and the Co-Ad group (Control over GSK1437173A + GSK2321138A) was below 1.5; Adjusted Geometric mean concentration ra = 1.08, 95% CI 2-sided [0.97 to 1.20]

4. Primary Outcome: FLU Haemagglutination Inhibition (HI) Antibody Titers
Description: For each strain included in the FLU-D-QIV vaccine, an ANOVA model was used to analyze post-vaccination log-transformed titers. The fixed-effect model included the minimization variable (age cohorts) and the treatment as fixed effect. The pre-vaccination log-transformed concentrations were included as continuous covariate. Geometric Means (GM) of post-vaccination titers (Day 21) were calculated conditionally to the means of the pre-vaccination log-transformed titers (Month 0) for each strain.
  Adjusted GMTs (GMTs adjusted for baseline titers) and Adjusted GMT ratios were calculated together with 2-sided 95% CIs.
Time Frame: At Day 21 post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 384 | 394
Titers
  Flu A/California/7/2009 H1N1 HI Day 21 | 187.5 [166.7 to 210.8] | 194.3 [173.0 to 218.1]
  Flu A/Texas/50/2012 H3N2 HI Day 21 | 63.7 [58.3 to 69.7] | 65.9 [60.3 to 72.0]
  Flu B/Brisbane/60/2008 Victoria HI Day 21 | 170.2 [156.1 to 185.6] | 181.6 [166.7 to 197.8]
  Flu B/Massachusetts/2/2012 Yamagata HI Day 21 | 423.5 [392.0 to 457.5] | 413.9 [383.4 to 446.8]
Statistical Analysis 1: Comparison: GSK1437173A + GSK2321138A Group vs Control Group; For the Flu A/California/7/2009 H1N1 strain ,an ANOVA model was used to analyze post-vaccination log-transformed titers. The fixed-effect model included the minimization variable (age cohorts) and the treatment as fixed effect. The pre-vaccination log-transformed concentrations were included as continuous covariate. GMs of post-vaccination titers (Day 21) were calculated conditionally to the means of the pre-vaccination log-transformed titers (Month 0) for this strain; Test type: Non-Inferiority or Equivalence — Comparisons at Day 21 after the FLU-D-QIV dose were performed between the Control group and GSK1437173A + GSK2321138A group. The GSK1437173A + GSK2321138A group was considered as statistically significant non inferior compared to the Control group in terms of immunogenicity (for each strain) if the UL of 2-sided 95% CI of the ratio of GMTs between the Control and the GSK1437173A + GSK2321138A (Control/ GSK1437173A + GSK2321138A) group is below 1.5; Adjusted geometric mean Titer ratio = 1.04, 95% CI 2-sided [0.88 to 1.22]
Statistical Analysis 2: Comparison: GSK1437173A + GSK2321138A Group vs Control Group; For the Flu A/Texas/50/2012 H3N2 strain ,an ANOVA model was used to analyze post-vaccination log-transformed titers. The fixed-effect model included the minimization variable (age cohorts) and the treatment as fixed effect. The pre-vaccination log-transformed concentrations were included as continuous covariate. GMs of post-vaccination titers (Day 21) were calculated conditionally to the means of the pre-vaccination log-transformed titers (Month 0) for this strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Adjusted geometric mean Titer ratio = 1.03, 95% CI 2-sided [0.91 to 1.17]
Statistical Analysis 3: Comparison: GSK1437173A + GSK2321138A Group vs Control Group; For the Flu B/Brisbane/60/2008 Victoria strain ,an ANOVA model was used to analyze post-vaccination log-transformed titers. The fixed-effect model included the minimization variable (age cohorts) and the treatment as fixed effect. The pre-vaccination log-transformed concentrations were included as continuous covariate. GMs of post-vaccination titers (Day 21) were calculated conditionally to the means of the pre-vaccination log-transformed titers (Month 0) for this strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Adjusted geometric mean Titer ratio = 1.07, 95% CI 2-sided [0.95 to 1.20]
Statistical Analysis 4: Comparison: GSK1437173A + GSK2321138A Group vs Control Group; For the Flu B/Massachusetts/2/2012 Yamagata strain ,an ANOVA model was used to analyze post-vaccination log-transformed titers. The fixed-effect model included the minimization variable (age cohorts) and the treatment as fixed effect. The pre-vaccination log-transformed concentrations were included as continuous covariate. GMs of post-vaccination titers (Day 21) were calculated conditionally to the means of the pre-vaccination log-transformed titers (Month 0) for this strain; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Adjusted geometric mean Titer ratio = 0.98, 95% CI 2-sided [0.88 to 1.09]

5. Secondary Outcome: Number of Subjects With FLU HI Antibody Titers ≥1:10
Description: FLU HI antibodies were assessed in four strains: Flu A/California/7/2009 H1N1, Flu A/Texas/50/2012 H3N2, Flu B/Brisbane/60/2008 Victoria and Flu B/Massachusetts (Massach)/2/2012 Yamagata (Yama). Cut-off titer for seropositivity was 1:10.
Time Frame: At Day 0 (PRE) and 21 post vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 386 | 395
Subjects
  Flu A/California/7/2009 H1N1 Day 0 [N=386,395] | 288 | 294
  Flu A/California/7/2009 H1N1Day 21 [N=384,394] | 381 | 389
  Flu A/Texas/50/2012 H3N2 Day 0 [N=386,395] | 283 | 300
  Flu A/Texas/50/2012 H3N2 Day 21 [N=384,394] | 380 | 392
  Flu B/Brisbane/60/2008 Victoria Day 0 [N=386,395] | 365 | 375
  Flu B/Brisbane/60/2008 Victoria Day 21 [N=384,394] | 383 | 394
  Flu B/Massach/2/2012 Yama Day 0 [N=386,395] | 376 | 389
  Flu B/Massach/2/2012 Yama Day21 [N=384,394] | 384 | 394

6. Secondary Outcome: Number of Seroprotected Subjects With HI Antibody Titers ≥ 1:40
Description: Seroprotection rate is defined as the percentage of vaccines with a serum HI titer ≥1:40 that usually was accepted as indicating protection. FLU HI antibodies were assessed in four strains: Flu A/California/7/2009 H1N1, Flu A/Texas/50/2012 H3N2, Flu B/Brisbane/60/2008 Victoria (Vic) and Flu B/Massachusetts(Massach)/2/2012 Yamagata (Yama).
Time Frame: At Day 0 (PRE) and at Day 21 post vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 386 | 395
Subjects
  Flu A/California/7/2009 H1N1 HI Day 0 [N=386,395] | 185 | 161
  Flu A/California/7/2009 H1N1 HI Day 21 [N=384,394] | 347 | 360
  Flu A/Texas/50/2012 H3N2 HI Day 0 [N=386,395] | 134 | 121
  Flu A/Texas/50/2012 H3N2 HI Day 21 [N=384,394] | 292 | 295
  Flu B/Brisbane/60/2008 Vic HI Day 0 [N=386,395] | 279 | 271
  Flu B/Brisbane/60/2008 Vic HI Day 21 [N=384,394] | 372 | 382
  Flu B/Massach/2/2012 Yama HI Day 0 [N=386,395] | 351 | 361
  Flu B/Massach/2/2012 Yama HI Day 21 [N=384,394] | 383 | 393

7. Secondary Outcome: FLU Haemagglutination Inhibition (HI) Antibody Titers
Description: HI antibody titres against the four influenza vaccine strains Flu A/California/7/2009, Flu A/Texas/50/2012, Flu B/Brisbane/60/2008 Victoria (Vic) and Flu B/Massachusetts (Massach)/2/2012 Yamagata (Yamma) were expressed as geometric mean titers (GMTs).
Time Frame: At Day 0 (PRE) and Day 21 post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 386 | 395
Titers
  Flu A/California/7/2009 H1N1 HI Day 0 [N=386,395] | 29 [25.1 to 33.5] | 24.9 [21.8 to 28.5]
  Flu A/California/7/2009 H1N1 HI Day 21[N=384,394] | 196.2 [172.2 to 223.5] | 193.2 [170.2 to 219.4]
  Flu A/Texas/50/2012 H3N2 HI Day 0 [N=386,395] | 19.6 [17.5 to 21.9] | 19.0 [17.1 to 21.1]
  Flu A/Texas/50/2012 H3N2 HI Day 21 [N=384,394] | 65.4 [59.0 to 72.5] | 66.8 [60.4 to 74.0]
  Flu B/Brisbane/60/2008 Vic HI Day 0 [N=386,395] | 52.2 [46.9 to 58.1] | 48.6 [43.7 to 54]
  Flu B/Brisbane/60/2008 Vic HI Day 21 [N=384,394] | 177.2 [161.6 to 194.2] | 185.2 [168 to 204.1]
  Flu B/Massach/2/2012 Yama HI Day 0 [N=386,395] | 128.8 [115.7 to 143.4] | 127 [114.9 to 140.3]
  Flu B/Massach/2/2012 Yama HI Day 21 [N=384,394] | 433.7 [401.3 to 468.7] | 423.3 [388 to 461.8]

8. Secondary Outcome: Number of Seroconverted Subjects in Terms of HI Antibodies
Description: The number of seroconverted subjects was assessed in terms of HI antibodies against the four influenza vaccine strains Flu A/California/7/2009, Flu A/Texas/50/2012, Flu B/Brisbane/60/2008 Victoria and Flu B/Massachusetts/2/2012 Yamagata.
Time Frame: At Day 21 post vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 384 | 394
Subjects
  Flu A/California/7/2009 H1N1 HI | 232 | 240
  Flu A/Texas/50/2012 H3N2 HI | 136 | 139
  Flu B/Brisbane/60/2008 Victoria HI | 143 | 169
  Flu B/Massachusetts/2/2012 Yamagata HI | 154 | 148

9. Secondary Outcome: Geometric Mean Ratio for Flu HI Antibodies Post-vaccination Titer
Description: The geometric mean ratio for Flu HI antibodies against the four influenza vaccine strains Flu A/California/7/2009, Flu A/Texas/50/2012, Flu B/Brisbane/60/2008 Victoria and Flu B/Massachusetts/2/2012 Yamagata was defined as the geometric mean of the within subject ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer.
Time Frame: At Day 21 post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 384 | 394
Ratio
  Flu A/California/7/2009 H1N1 HI | 6.8 [5.9 to 7.8] | 7.7 [6.7 to 9]
  Flu A/Texas/50/2012 H3N2 HI | 3.4 [3.0 to 3.7] | 3.5 [3.2 to 4.0]
  Flu B/Brisbane/60/2008 Victoria HI | 3.4 [3 to 3.8] | 3.8 [3.4 to 4.3]
  Flu B/Massachusetts/2/2012 Yamagata HI | 3.4 [3 to 3.7] | 3.3 [3 to 3.7]

10. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 (G3) pain = pain that prevented normal activity. Grade 3 (G3) redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: Within 7 days (Days 0-6) after each vaccine dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered, on subjects with their symptom sheets completed.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 410 | 412
Subjects
  Any Pain D1 GSK 2321138A [N=410;412] | 140 | 112
  G3 Pain D1 GSK 2321138A [N=410;412] | 7 | 4
  Any Redness D1 GSK 2321138A [N=410;412] | 31 | 37
  G3 Redness D1 GSK 2321138A [N=410;412] | 1 | 2
  Any Swelling D1 GSK 2321138A [N=410;412] | 16 | 18
  G3 Swelling D1 GSK 2321138A [N=410;412] | 0 | 1
  Any Pain D2 GSK 2321138A [N=0;0] | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP
  G3 Pain D2 GSK 2321138A [N=0;0] | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP
  Any Redness D2 GSK 2321138A [N=0;0] | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP
  G3 Redness D2 GSK 2321138A [N=0;0] | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP
  Any Swelling D2 GSK 2321138A [N=0;0] | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP
  G3 Swelling D2 GSK 2321138A [N=0;0] | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A GROUP
  Any Pain D1 GSK 1437173A [N=410;0] | 292 | NA — No data was available for the GSK 1437173A vaccine at Dose 1 for the Control Group, as it was only administered at Doses 2 and 3 in this group.
  G3 Pain D1 GSK 1437173A [N=410;0] | 31 | NA — No data was available for the GSK 1437173A vaccine at Dose 1 for the Control Group, as it was only administered at Doses 2 and 3 in this group.
  Any Redness D1 GSK 1437173A [N=410;0] | 112 | NA — No data was available for the GSK 1437173A vaccine at Dose 1 for the Control Group, as it was only administered at Doses 2 and 3 in this group.
  G3 Redness D1 GSK 1437173A [N=410;0] | 4 | NA — No data was available for the GSK 1437173A vaccine at Dose 1 for the Control Group, as it was only administered at Doses 2 and 3 in this group.
  Any Swelling D1 GSK 1437173A [N=410;0] | 64 | NA — No data was available for the GSK 1437173A vaccine at Dose 1 for the Control Group, as it was only administered at Doses 2 and 3 in this group.
  G3 Swelling D1 GSK 1437173A [N=410;0] | 0 | NA — No data was available for the GSK 1437173A vaccine at Dose 1 for the Control Group, as it was only administered at Doses 2 and 3 in this group.
  Any Pain D2 GSK 1437173A [N=403;405] | 290 | 280
  G3 Pain D2 GSK 1437173A [N=403;405] | 32 | 25
  Any Redness D2 GSK 1437173A [N=403;405] | 103 | 91
  G3 Redness D2 GSK 1437173A [N=403;405] | 5 | 6
  Any Swelling D2 GSK 1437173A [N=403;405] | 64 | 47
  G3 Swelling D2 GSK 1437173A [N=403;405] | 0 | 0
  Any Pain D3 GSK 2321138A [N=0;0] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A
  G3 Pain D3 GSK 2321138A [N=0;0] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A
  Any Redness D3 GSK 2321138A [N=0;0] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A
  G3 Redness D3 GSK 2321138A [N=0;0] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A
  Any Swelling D3 GSK 2321138A [N=0;0] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A
  G3 Swelling D3 GSK 2321138A [N=0;0] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | NA — No data was available for the GSK2321138A vaccine at Doses 2 and 3 for any of the groups, as it was only administered at Dose 1 for the GSK1437173A + GSK2321138A
  Any Pain D3 GSK 1437173A [N=0;402] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | 269
  G3 Pain D3 GSK 1437173A [N=0;402] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | 25
  Any Redness D3 GSK 1437173A [N=0;402] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | 100
  G3 Redness D3 GSK 1437173A [N=0;402] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | 7
  Any Swelling D3 GSK 1437173A [N=0;402] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | 50
  G3 Swelling D2 GSK 1437173A [N=0;402] | NA — No data was available for the GSK1437173A + GSK2321138A GROUP at Dose 3, since it only received 2 vaccine doses. | 4

11. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: Within 7 days (Days 0-6) across doses
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 411 | 413
Subjects
  Any Pain Across Doses | 344 | 318
  Grade 3 Pain Across Doses | 55 | 40
  Any Redness Across Doses | 153 | 144
  Grade 3 Redness Across Doses | 9 | 14
  Any Swelling Across Doses | 99 | 86
  Grade 3 Swelling Across Doses | 0 | 5

12. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 7 days (Days 0-6) after each vaccine dose
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group
Number analyzed (Participants) | 409
Subjects
  Any Arthralgia Dose 1 [N=409] | 89
  Grade 3 Arthralgia Dose 1 [N=409] | 8
  Related Arthralgia Dose 1 [N=409] | 67
  Any Fatigue Dose 1 [N=409] | 150
  Grade 3 Fatigue Dose 1 [N=409] | 15
  Related Fatigue Dose 1 [N=409] | 107
  Any Gastrointestinal Dose 1 [N=409] | 57
  Grade 3 Gastrointestinal Dose 1 [N=409] | 5
  Related Gastrointestinal Dose 1 [N=409] | 28
  Any Headache Dose 1 [N=409] | 122
  Grade 3 Headache Dose 1 [N=409] | 5
  Related Headache Dose 1 [N=409] | 80
  Any Myalgia Dose 1 [N=409] | 135
  Grade 3 Myalgia Dose 1 [N=409] | 11
  Related Myalgia Dose 1 [N=409] | 105
  Any Shivering Dose 1 [N=409] | 101
  Grade 3 Shivering Dose 1 [N=409] | 12
  Related Shivering Dose 1 [N=409] | 86
  Any Temperature Dose 1 [N=409] | 63
  Grade 3 Temperature Dose 1 [N=409] | 1
  Related Temperature Dose 1 [N=409] | 53
  Any Arthralgia Dose 2 [N=402] | 114
  Grade 3 Arthralgia Dose 2 [N=402] | 16
  Related Arthralgia Dose 2 [N=402] | 94
  Any Fatigue Dose 2 [N=402] | 167
  Grade 3 Fatigue Dose 2 [N=402] | 23
  Related Fatigue Dose 2 [N=402] | 138
  Any Gastrointestinal Dose 2 [N=402] | 47
  Grade 3 Gastrointestinal Dose 2 [N=402] | 3
  Related Gastrointestinal Dose 2 [N=402] | 32
  Any Headache Dose 2 [N=402] | 136
  Grade 3 Headache Dose 2 [N=402] | 16
  Related Headache Dose 2 [N=402] | 109
  Any Myalgia Dose 2 [N=402] | 157
  Grade 3 Myalgia Dose 2 [N=402] | 18
  Related Myalgia Dose 2 [N=402] | 135
  Any Shivering Dose 2 [N=402] | 142
  Grade 3 Shivering Dose 2 [N=402] | 30
  Related Shivering Dose 2 [N=402] | 122
  Any Temperature Dose 2 [N=402] | 74
  Grade 3 Temperature Dose 2 [N=402] | 1
  Related Temperature Dose 2 [N=402] | 63

13. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 12
Time Frame: Within 7 days (Days 0-6) after each vaccine dose
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Control Group
Number analyzed (Participants) | 411
Subjects
  Any Arthralgia, Dose 1 [N=411] | 37
  Grade 3 Arthralgia, Dose 1 [N=411] | 8
  Related Arthralgia, Dose 1 [N=411] | 25
  Any Fatigue, Dose 1 [N=411] | 52
  Grade 3 Fatigue, Dose 1 [N=411] | 4
  Related Fatigue, Dose 1 [N=411] | 33
  Any Gastrointestinal, Dose 1 [N=411] | 32
  Grade 3 Gastrointestinal, Dose 1 [N=411] | 2
  Related Gastrointestinal, Dose 1 [N=411] | 16
  Any Headache, Dose 1 [N=411] | 57
  Grade 3 Headache, Dose 1 [N=411] | 2
  Related Headache, Dose 1 [N=411] | 31
  Any Myalgia, Dose 1 [N=411] | 55
  Grade 3 Myalgia, Dose 1 [N=411] | 4
  Related Myalgia, Dose 1 [N=411] | 45
  Any Shivering, Dose 1 [N=411] | 30
  Grade 3 Shivering, Dose 1 [N=411] | 0
  Related Shivering, Dose 1 [N=411] | 25
  Any Temperature, Dose 1 [N=411] | 18
  Grade 3 Temperature, Dose 1 [N=411] | 0
  Related Temperature, Dose 1 [N=411] | 15
  Any Arthralgia, Dose 2 [N=405] | 67
  Grade 3 Arthralgia, Dose 2 [N=405] | 6
  Related Arthralgia, Dose 2 [N=405] | 51
  Any Fatigue, Dose 2 [N=405] | 108
  Grade 3 Fatigue, Dose 2 [N=405] | 9
  Related Fatigue, Dose 2 [N=405] | 87
  Any Gastrointestinal, Dose 2 [N=405] | 37
  Grade 3 Gastrointestinal, Dose 2 [N=405] | 1
  Related Gastrointestinal, Dose 2 [N=405] | 28
  Any Headache, Dose 2 [N=405] | 87
  Grade 3 Headache, Dose 2 [N=405] | 8
  Related Headache, Dose 2 [N=405] | 70
  Any Myalgia, Dose 2 [N=405] | 135
  Grade 3 Myalgia, Dose 2 [N=405] | 7
  Related Myalgia, Dose 2 [N=405] | 115
  Any Shivering, Dose 2 [N=405] | 87
  Grade 3 Shivering, Dose 2 [N=405] | 10
  Related Shivering, Dose 2 [N=405] | 75
  Any Temperature, Dose 2 [N=405] | 44
  Grade 3 Temperature, Dose 2 [N=405] | 1
  Related Temperature, Dose 2 [N=405] | 34
  Any Arthralgia, Dose 3 [N=402] | 95
  Grade 3 Arthralgia, Dose 3 [N=402] | 18
  Related Arthralgia, Dose 3 [N=402] | 79
  Any Fatigue, Dose 3 [N=402] | 149
  Grade 3 Fatigue, Dose 3 [N=402] | 31
  Related Fatigue, Dose 3 [N=402] | 120
  Any Gastrointestinal, Dose 3 [N=402] | 63
  Grade 3 Gastrointestinal, Dose 3 [N=402] | 6
  Related Gastrointestinal, Dose 3 [N=402] | 46
  Any Headache, Dose 3 [N=402] | 133
  Grade 3 Headache, Dose 3 [N=402] | 23
  Related Headache, Dose 3 [N=402] | 111
  Any Myalgia, Dose 3 [N=402] | 138
  Grade 3 Myalgia, Dose 3 [N=402] | 24
  Related Myalgia, Dose 3 [N=402] | 121
  Any Shivering, Dose 3 [N=402] | 147
  Grade 3 Shivering, Dose 3 [N=402] | 23
  Related Shivering, Dose 3 [N=402] | 131
  Any Temperature, Dose 3 [N=402] | 87
  Grade 3 Temperature, Dose 3 [N=402] | 2
  Related Temperature, Dose 3 [N=402] | 70

14. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: as for outcome 12
Time Frame: Within 7 days (Days 0-6) across doses
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 411 | 413
Subjects
  Any Arthralgia, Across Doses | 154 | 135
  Grade 3 Arthralgia, Across Doses | 23 | 24
  Related Arthralgia, Across Doses | 121 | 110
  Any Fatigue, Across Doses | 224 | 186
  Grade 3 Fatigue, Across Doses | 30 | 38
  Related Fatigue, Across Doses | 175 | 151
  Any Gastrointestinal, Across Doses | 90 | 92
  Grade 3 Gastrointestinal, Across Doses | 6 | 9
  Related Gastrointestinal, Across Doses | 49 | 66
  Any Headache, Across Doses | 183 | 170
  Grade 3 Headache, Across Doses | 20 | 28
  Related Headache, Across Doses | 140 | 142
  Any Myalgia, Across Doses | 201 | 201
  Grade 3 Myalgia, Across Doses | 27 | 30
  Related Myalgia, Across Doses | 167 | 177
  Any Shivering, Across Doses | 174 | 181
  Grade 3 Shivering, Across Doses | 35 | 30
  Related Shivering, Across Doses | 151 | 159
  Any Temperature, Across Doses | 107 | 119
  Grade 3 Temperature, Across Doses | 2 | 3
  Related Temperature, Across Doses | 90 | 96

15. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During 30 days (Days 0-29) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 413 | 415
Subjects
  Any AEs | 110 | 162
  Grade 3 AEs | 17 | 29
  Related AEs | 18 | 26

16. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From first vaccination up to Month 18 (study end)
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 413 | 415
Subjects | 42 | 39

17. Secondary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination up to Month 18 (study end)
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Number analyzed (Participants) | 413 | 415
Subjects | 4 | 2

ADVERSE EVENTS:
Time Frame: Systematically-assessed symptoms: Days 0-7 post each vaccine dose; AEs: Days 0-29 post each vaccine dose; SAEs: from Day 0 to Month 18
Description: There were shifts in the total SAE numbers: GSK1437173A + GSK2321138A Group: 1 subject whose myasthenia gravis (initially not reported as SAE) became an SAE at the final analysis; The Psychotic disorder was renamed Depression; Control Group: initial worsening of hiatal hernia for 1 was later not considered an SAE.
Arm/Group | GSK1437173A + GSK2321138A Group | Control Group
Serious Adverse Events (participants affected / at risk) | 42/413 | 39/415
Other Adverse Events (participants affected / at risk) | 370/413 | 369/415
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1437173A + GSK2321138A Group (N=413) | Control Group (N=415)
Coronary artery disease (Cardiac disorders) | 3 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Hypertension (Vascular disorders) | 1 | 2
Pneumonia (Infections and infestations) | 3 | 0
Syncope (Nervous system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 2 | 0
Acquired syringomyelia (Nervous system disorders) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Asthenia (General disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis pharyngeal (Infections and infestations) | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Occipital neuralgia (Nervous system disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Transitional cell carcinoma (Nervous system disorders) | 1 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Death (unknown causes) (General disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK1437173A + GSK2321138A Group (N=413) | Control Group (N=415)
Nasopharyngitis (Infections and infestations) | 14 | 22
Pain (General disorders) | 344/411 | 318/413
Redness (General disorders) | 153/411 | 144/413
Swelling (General disorders) | 99/411 | 86/413
Arthralgia (General disorders) | 154/411 | 135/413
Fatigue (General disorders) | 224/411 | 186/413
Gastrointestinal (General disorders) | 90/411 | 92/413
Headache (General disorders) | 183/411 | 170/413
Myalgia (General disorders) | 201/411 | 201/413
Shivering (General disorders) | 174/411 | 181/413
Temperature/(Oral) (General disorders) | 107/411 | 119/413

LIMITATIONS AND CAVEATS:
The current data reflect the data reported in the database at the time of the end-of-study analysis. The previous data were based on the primary analysis including a safety analysis up to the data lock point of 7-APR-2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.